CLINICAL TRIAL: NCT00766025
Title: A Phase I, Open Label, Parallel Group, Single and Multiple Dose Study in Taiwanese Subjects Identified as CYP2C19 Poor Metabolizers or Extensive Metabolizers Receiving 20 Milligrams of Rosuvastatin Calcium
Brief Title: Study in Taiwanese Subjects Identified as CYP2C19 Poor and Extensive Metabolizers Receiving Rosuvastatin
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Michael Cressman, Medical Science Executive Director, Clinical Development, Cardiovascular, AstraZeneca Pharmaceuticals
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: D3560C00059; Rosuvastatin Calcium
Record Dates: First submitted 2008-10-02; First posted 2008-10-03 (Estimated); Last update posted 2009-03-02 (Estimated); Status verified 2009-02

CONDITIONS: CYP2C19 Poor; Extensive Metabolizers
Keywords: Taiwanese Subjects; CYP2C19; Poor Metabolizers; Extensive Metabolizers; Taiwanese Subjects identified as CYP2C19 Poor or Extensive Metabolizers
MeSH Terms: interventions — Rosuvastatin Calcium

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Rosuvastatin Calcium (Experimental)
  Interventions: Drug: Rosuvastatin Calcium

INTERVENTIONS:
Drug: Rosuvastatin Calcium — single oral dose on days 1, 4, 5, 6, 10-16, 17

SUMMARY:
The main purpose of this study is to examine Taiwanese subjects identified as CYP2C19 poor and extensive metabolizers while taking single and multiple dosing a rosuvastatin calcium.

ELIGIBILITY:
Inclusion Criteria:

* Subject must have blood drawn for genotyping (determination of EM or PM of CYP2C19, determination of OATP-C1B1, BCRP 421C>A, and CYP2C9.
* Males and females aged 20-65, inclusive
* Women who are surgically sterilized, post-menopausal for at least one year, or not pregnant and/or lactating. Women of childbearing potential must be willing to abstain from sexual activity or use an effective contraception as outlined in protocol.

Exclusion Criteria:

* Subjects with deoxyribonucleic acid (DNA) that codes for OATP-C 1B1 *5 and *15, BCRP 421C>A and/or non wild-type CYP2C9
* History of adverse drug reaction or hypersensitivity to statins or drugs with a similar chemical structure to rosuvastatin
* History or presence of gastrointestinal, hepatic, or renal disease or other conditions known to interfere with absorption, distribution, metabolism and excretion (ADME) of drugs
* Any contraindication determined by review of a detailed medical and drug history, complete physical examination, vital signs, blood chemistry, hematology, and electrocardiogram (ECG)

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2008-09; Study Completion 2009-02 (Actual)

PRIMARY OUTCOMES:
Blood levels of rosuvastatin in Taiwanese subjects identified as CYP2CIP poor and extensive metabolizers | Scheduled times during the 18 days that the study drug is taken
Blood levels for assessment of pharmacodynamic (lipid) parameters | Days -1 and 18

SECONDARY OUTCOMES:
Safety and tolerability of rosuvastatin in Taiwanese subjects identified as CYP2C19 poor and extensive metabolizers | Screening through completion of the study

CONTACTS AND LOCATIONS:
Overall Officials: Regeio Mosquea-Garcia, MD, Study Director — AstraZeneca; Robin Meng, MD, PhD, Study Director — AstraZeneca; Tzung-Dau Wang, MD, Principal Investigator — Northern Taiwan University Hospital
Locations (1):
- Research Site, Taipei, Taiwan